CLINICAL TRIAL: NCT00567164
Title: A Multicenter, Open-label, Three-arm, Active-controlled Study to Assess the Efficacy and Safety of the Oral Contraceptive SH T00186D (0.02 mg Ethinyl Estradiol as Betadex Clathrate and 3 mg Drospirenone) in Two Flexible Extended Regimens and a Conventional Regimen of YAZ in 1756 Healthy Females for 1 Year
Brief Title: Efficacy and Safety of Two Flexible Extended Regimens of BAY86-5300 (SH T00186D) in Comparison With the Conventional Regimen of YAZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91698; 311642 (Other: Bayer)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-01

CONDITIONS: Contraception; Ovulation Inhibition; Contraceptives, Oral
Keywords: Oral Contraception; Birth Control pill; Healthy women requesting oral contraception; Contraceptive efficacy
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Flexible (extended) regimen no. 1 of EE20/DRSP (BAY86-5300) (Experimental): Minimum of 3 cycles of treatment, each cycle comprising 120 days (maximum) intended treatment with one tablet daily of BAY86-5300 (SH T00186D) followed by a 4-day tablet-free interval. If 3 consecutive days of bleeding and/or spotting occurred between days 25 to 120 of the treatment cycle, a 4-day tablet-free interval was advised. The minimum period between 2 tablet-free intervals was 24 days. After each 4-day tablet-free interval, a new 124-day intended treatment cycle was to be restarted, resulting in a minimum of 3 and maximum of 13 withdrawal bleeding episodes during one year of treatment
  Interventions: Drug: EE20/DRSP (BAY86-5300)
- Flexible (extended) regimen no. 2 of EE20/DRSP (BAY86-5300) (Experimental): Minimum of 3 cycles of treatment, each cycle comprising 120 days (maximum) uninterrupted treatment with one tablet daily of BAY86-5300 (SH T00186D) and a 4-day tablet-free interval. Subjects were permitted to schedule their withdrawal bleeding (ie, 4-day tablet-free interval) at any time between days 25 to 120 of the cycle. Subjects had the option to follow the bleeding rules of the flexible (extended) regimen no. 1 of BAY86-5300. The minimum period between 2 tablet-free intervals was 24 days. After each 4-day tablet-free interval, a new 124-day intended treatment cycle was to be restarted, resulting in a minimum of 3 and maximum of 13 withdrawal bleeding episodes during one year of treatment.
  Interventions: Drug: EE20/DRSP (BAY86-5300)
- Conventional regimen of EE20/DRSP (YAZ, BAY86-5300) (Active Comparator): 13 cycles of treatment, each cycle comprising an intake of one tablet daily with 24 days of active tablets of BAY86-5300 (YAZ, SH T00186D) followed by 4 days of tablets without active substance (together resulting in one cycle of 24+4 standard treatment). 13 withdrawal bleeding episodes during one year of treatment were expected.
  Interventions: Drug: EE20/DRSP (YAZ, BAY86-5300)

INTERVENTIONS:
Drug: EE20/DRSP (BAY86-5300) — Combination tablet containing 0.02 mg ethinyl estradiol as betadex clathrate and 3.0 mg drospirenone
  Other Names: SH T00186D
  Arms: Flexible (extended) regimen no. 1 of EE20/DRSP (BAY86-5300)
Drug: EE20/DRSP (BAY86-5300) — Combination tablet containing 0.02 mg ethinyl estradiol as betadex clathrate and 3.0 mg drospirenone
  Other Names: SH T00186D
  Arms: Flexible (extended) regimen no. 2 of EE20/DRSP (BAY86-5300)
Drug: EE20/DRSP (YAZ, BAY86-5300) — Fixed package per cycle containing combination tablets containing 0.02 mg ethinyl estradiol as betadex clathrate and 3.0 mg drospirenone (24 per cycle) + tablets without active substance (4 per cycle)
  Other Names: SH T00186D
  Arms: Conventional regimen of EE20/DRSP (YAZ, BAY86-5300)

SUMMARY:
The purpose of this study is to determine whether the study drug is safe and effective.

DETAILED DESCRIPTION:
The primary efficacy parameter is the number of observed unintended pregnancy during 1 year of treatment. Secondary efficacy parameter include bleeding parameters and menstrual related symptoms Safety parameters included assessment of adverse events, laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

- Healthy women between 18 and 45 requesting oral contraception. Smokers may not exceed 35 years of age.

Exclusion Criteria:

- The use of steroidal oral contraceptives, or any drug that could alter oral contraception metabolism will be prohibited during the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1887 (Actual)
Dates: Start 2007-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (77):
- United States (77):
  - Montgomery, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Beverly Hills, California
  - Pacific Palisades, California
  - San Diego, California
  - Santa Ana, California
  - Vallejo, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Greenwood Village, Colorado
  - Littleton, Colorado
  - Waterbury, Connecticut
  - Boynton Beach, Florida
  - Brooksville, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Crystal River, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - Naples, Florida
  - North Miami, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Champaign, Illinois
  - Chicago, Illinois
  - Newburgh, Indiana
  - Wichita, Kansas
  - Lexington, Kentucky
  - Marrero, Louisiana
  - Paw Paw, Michigan
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - LasVegas, Nevada
  - Moorestown, New Jersey
  - New Brunswick, New Jersey
  - Rochester, New York
  - Durham, North Carolina
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Mt. Pleasant, South Carolina
  - Chattanooga, Tennessee
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Colleyville, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - West Jordan, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- [Result] Jensen JT, Garie SG, Trummer D, Elliesen J. Bleeding profile of a flexible extended regimen of ethinylestradiol/drospirenone in US women: an open-label, three-arm, active-controlled, multicenter study. Contraception. 2012 Aug;86(2):110-8. doi: 10.1016/j.contraception.2011.12.009. Epub 2012 Jan 26. PMID 22281416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of first subject, first visit was 22 Oct 2007. The date of last subject, last visit was 11 Nov 2009.
Pre-assignment Details: A total of 2450 subjects were screened ; 563 failed screening. The remaining 1887 subjects were assigned to treatment. Of these, 1864 (98.8%) were in the Full Analysis Set (FAS), ie, study medication was dispensed to them and they had at least 1 post-baseline observation. A total of 1196 (63.4%) subjects completed the study.
Groups:
- Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300): 13 cycles of treatment, each cycle comprising an intake of one tablet daily with 24 days of active tablets of BAY86-5300 (YAZ, SH T00186D) followed by 4 days of placebo tablets (SH T470PD). 13 withdrawal bleeding episodes during one year of treatment were expected.
Period: Overall Study
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Started | 1421 | 234 | 232
Subjects Received Treatment | 1406 (Full Analysis Set) | 232 (Full Analysis Set) | 226 (Full Analysis Set)
Completed | 875 | 161 | 160
Not Completed | 546 | 73 | 72
Not completed — Withdrawal by Subject | 171 | 21 | 17
Not completed — Protocol Violation | 23 | 4 | 2
Not completed — Adverse Event | 92 | 13 | 9
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 202 | 23 | 21
Not completed — Pregnancy | 20 | 4 | 6
Not completed — Primary Reason coded as 'Other' | 37 | 8 | 16
Not completed — Missing | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300) | Total
Number analyzed (Participants) | 1406 | 232 | 226 | 1864
Age, Continuous [Mean (Standard Deviation); unit: years] — Only describes treated participants
  years | 25.2 (4.5) | 26.8 (6.8) | 27.3 (6.4) | 25.7 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Only describes treated participants
  Participants
    Female | 1406 | 232 | 226 | 1864
    Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pearl Index
Description: The Pearl Index (PI) is the number of pregnancies per 100 woman years. The PI is obtained by dividing the number of pregnancies during treatment (conception date on/after the 1st day of treatment and not later than last day of treatment +14 days) by the treatment exposure time (in 100 women years) that the women were under risk of getting pregnant. The Pearl Index was not calculated individually for either the Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) treatment arm, nor for the Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300) treatment arm, because the low sample size in these treatment arms (approximately. 200 subjects per group) did not allow a reliable PI calculation of these groups alone.
Time Frame: Up to 1 year
Population: Full Analysis Set of Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) treatment arm. Pooled Full Analysis Sets of Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) and Regimen no. 2 of EE20/DRSP (BAY86-5300) treatment arms.
Measure: Mean (95% Confidence Interval); unit: Pregnancies per 100 years of exposure
Groups:
- Pooled Analysis of Flexible Regimen no. 1 and Regimen no. 2: Pooled FAS of Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) (see first arm) and Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300). Regimen no. 2: Minimum of 3 cycles of treatment, each cycle comprising 120 days (maximum) uninterrupted treatment with one tablet daily of BAY86-5300 (SH T00186D) and a 4-day tablet-free interval. Subjects were permitted to schedule their withdrawal bleeding (ie, 4-day tablet-free interval) at any time between days 25 to 120 of the cycle. Subjects had the option to follow the bleeding rules of the flexible (extended) regimen no. 1 of BAY86-5300. The minimum period between 2 tablet-free intervals was 24 days. After each 4-day tablet-free interval, a new 124-day intended treatment cycle was to be restarted, resulting in a minimum of 3 and maximum of 13 withdrawal bleeding episodes during one year of treatment.
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Pooled Analysis of Flexible Regimen no. 1 and Regimen no. 2
Number analyzed (Participants) | 1406 | 1638
Pregnancies per 100 years of exposure | 1.65 [0.96 to 2.65] | 1.92 [1.22 to 2.89]

2. Secondary Outcome: Number of Bleeding Days (Including Spotting Days)
Description: Number of days per participant with bleeding or spotting
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1317 | 222 | 207
Days | 39.9 (29.6) | 46.8 (33.1) | 51.8 (34.6)
Statistical Analysis 1: Comparison: Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) vs Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300); Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -11.85, 95% CI [-16.3 to -7.394], Standard Deviation 30.356

3. Secondary Outcome: Number of Bleeding Days (Excluding Spotting Days)
Description: Number of days per participant with bleeding (excluding spotting days)
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1317 | 222 | 207
Days | 19.4 (15.7) | 21.4 (15.6) | 32.9 (23.5)

4. Secondary Outcome: Number of Days With Bleeding (Including and Excluding Spotting) Within 90-day Reference Period 1.
Description: Number of days per participant with bleeding (including and excluding spotting) within 90-day reference period 1. Reference period 1 (Day 1 to Day 90) was a 90 day period starting with the initial intake of study medication (protocol-specified to occur on first day of menstrual or withdrawal bleeding after screening). Therefore, the first 90-day reference period contains additional bleeding days (associated with the menstrual cycle prior to the start of study medication) when compared to any other reference period.
Time Frame: Day 1 to Day 90
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for reference period 1.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1067 | 176 | 169
Days
  Including days with spotting | 16.6 (12.2) | 18.5 (12.9) | 19.7 (9.8)
  Excluding days with spotting | 8.3 (6.9) | 9.1 (7.2) | 12.6 (6.5)

5. Secondary Outcome: Number of Days With Bleeding (Including and Excluding Spotting) Within 90-day Reference Period 2.
Description: Number of days per participant with bleeding (including and excluding spotting) within 90-day reference period 2. Reference period 2 (Day 91 to Day 180) was a 90-day period that started with the intake of study medication at the beginning of Cycle 4.
Time Frame: Day 91 to Day 180
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for reference period 2.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 950 | 161 | 145
Days
  Including days with spotting | 11.0 (9.7) | 12.5 (10.5) | 14.8 (8.0)
  Excluding days with spotting | 5.1 (5.2) | 5.4 (5.5) | 9.7 (6.3)

6. Secondary Outcome: Number of Days With Bleeding (Including and Excluding Spotting) Within 90-day Reference Period 3
Description: Number of days per participant with bleeding (including and excluding spotting) within 90-day reference period 3. Reference period 3 (Day 181 to Day 270) was a 90-day period that started with the intake of study medication at the beginning of Cycle 7.
Time Frame: Day 181 to Day 270
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for reference period 3.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 863 | 156 | 131
Days
  Including days with spotting | 10.0 (8.7) | 11.4 (10.8) | 14.8 (8.0)
  Excluding days with spotting | 4.7 (4.8) | 4.9 (5.0) | 9.4 (6.5)

7. Secondary Outcome: Number of Days With Bleeding/ (Including and Excluding Spotting) Within 90-day Reference Period 4
Description: Number of days per participant with bleeding (including and excluding spotting) within 90-day reference period 4. Reference period 4 (Day 271 to Day 360) was a 90-day period that started with the intake of study medication at the beginning of Cycle 10.
Time Frame: Day 271 to Day 360
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for reference period 4.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 808 | 143 | 112
Days
  Including days with spotting | 9.0 (9.2) | 9.5 (10.3) | 13.6 (7.3)
  Excluding days with spotting | 4.2 (4.8) | 4.0 (4.8) | 8.4 (5.5)

8. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 1
Description: A withdrawal bleeding episode (WBE) for the two flexible (extended) treatment arms 1) Ended at the earliest 4 days before the first day of the pill break of that cycle or later, AND 2) Started before or at the latest on the 4th day of the next cycle. For the conventional 24+4 treatment arm, a WBE 1) Started on or after Day 21 of that cycle, and lasted at least until Day 25 of the same cycle, OR 2) Started on or after Day 25 of that cycle, but before Day 25 of the next cycle. If more than one episode satisfied the above criteria, the first episode to occur was considered to be the WBE.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1124 | 191 | 187
Percentage of Participants | 84.2 | 83.8 | 66.8

9. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 2
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 2.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1025 | 176 | 180
Percentage of Participants | 85.9 | 84.7 | 86.7

10. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 3
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 3.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 868 | 154 | 182
Percentage of Participants | 78.6 | 79.2 | 84.6

11. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 4
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 4.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 601 | 121 | 161
Percentage of Participants | 73.4 | 66.1 | 86.3

12. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 5
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 5.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 368 | 71 | 155
Percentage of Participants | 78.0 | 69.0 | 85.8

13. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 6
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 6.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 229 | 43 | 155
Percentage of Participants | 77.7 | 69.8 | 85.2

14. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 7
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 7.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 129 | 30 | 144
Percentage of Participants | 78.3 | 70.0 | 84.0

15. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 8
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 8.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 78 | 13 | 143
Percentage of Participants | 82.1 | 69.2 | 86.7

16. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 9
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 9.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 46 | 10 | 138
Percentage of Participants | 73.9 | 80.0 | 85.5

17. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 10
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 10.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 19 | 10 | 130
Percentage of Participants | 78.9 | 70.0 | 84.6

18. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 11
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 11.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 9 | 8 | 128
Percentage of Participants | 55.6 | 62.5 | 85.9

19. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 12
Description: as for outcome 8
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 4 | 3 | 117
Percentage of Participants | 0 | 33.3 | 78.6

20. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 13
Description: A withdrawal bleeding episode (WBE) for the two flexible (extended) treatment arms 1) Ended at the earliest 4 days before the first day of the pill break of that cycle or later, AND 2) Started before or at the latest on the 4th day of the next cycle. For the conventional 24+4 treatment arm, a WBE 1) Started on or after Day 21 of that cycle, and lasted at least until Day 25 of the same cycle, OR 2) Started on or after Day 25 of that cycle, but before Day 25 of the next cycle. If more than one episode satisfied the above criteria, the first episode to occur was considered to be the WBE. There were no participants who provided bleeding data for cycle 13 in the Flexible (extended) regimen no.1 of EE20/DRSP (BAY86-5300), although one women did receive 13 cycles of treatment.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 13.
Measure: Number; unit: Percentage of Participants
Arm/Group | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1 | 73
Percentage of Participants | 0 | 20.5

21. Secondary Outcome: Percentage of Participants With a Withdrawal Bleeding Episode for Cycle 14
Description: A withdrawal bleeding episode (WBE) for the two flexible (extended) treatment arms 1) Ended at the earliest 4 days before the first day of the pill break of that cycle or later, AND 2) Started before or at the latest on the 4th day of the next cycle. For the conventional 24+4 treatment arm, a WBE 1) Started on or after Day 21 of that cycle, and lasted at least until Day 25 of the same cycle, OR 2) Started on or after Day 25 of that cycle, but before Day 25 of the next cycle. If more than one episode satisfied the above criteria, the first episode to occur was considered to be the WBE. There were no participants who received treatment in cycle 14 in the Flexible (extended) regimen no.1 of EE20/DRSP (BAY86-5300). There were no participants who provided bleeding data for cycle 14 in the Flexible (extended) regimen no.2 of EE20/DRSP (BAY86-5300), although one woman did receive 14 cycles of treatment.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding data for cycle 14.
Measure: Number; unit: Percentage of Participants
Arm/Group | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 11
Percentage of Participants | 9.1

22. Secondary Outcome: Number of Intracyclic Bleeding Days
Description: Intracyclic bleeding was considered any bleeding/spotting that occurred between withdrawal bleedings.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding and tablet intake data sufficient to calculate intracyclic bleeding.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1222 | 208 | 201
Days
  Including spotting only episodes | 8.0 (11.8) | 14.4 (19.1) | 7.1 (12.7)
  Excluding spotting only episodes | 3.6 (7.9) | 7.3 (12.8) | 5.2 (11.4)

23. Secondary Outcome: Number of Scheduled and Unscheduled Bleeding Days
Description: Scheduled bleeding is any bleeding/spotting (bl/sp) that occurs during the tablet free interval through the next 4 days of the subsequent treatment cycle. Unscheduled bleeding is any bl/sp that occurs while taking active hormones, except for bl/sp that occurs during the tablet free interval through day 4 of the subsequent treatment cycle or bl/sp on days 1-7 of treatment cycle 1.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). The number of participants analyzed only includes women who provided bleeding and tablet intake data sufficient to calculate scheduled/unscheduled bleeding. Analysis was only performed for the flexible and stop-and-go extended regimens.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300)
Number analyzed (Participants) | 1316 | 222
Days
  Scheduled bleeding days | 20.6 (14.1) | 21.9 (13.9)
  Unscheduled bleeding days | 20.0 (20.4) | 25.3 (27.8)

24. Secondary Outcome: Length of Cycles
Description: Cycle length per cycle. For the flexible and stop and go extended treatment arms, a treatment cycle started with the first day of pill intake after a tablet-free interval and ended with the last day of the subsequent tablet-free interval. A tablet-free interval (treatment withdrawal) was defined as at least 3 consecutive days without tablet intake. For the standard 24+4 treatment arm, a new cycle started each time a new blister pack of medication was started.
Time Frame: Up to 1 year
Population: Full Analysis Set (ie, all treated participants). Only cycle data from participants with sufficient data to calculate cycle length are included.
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Cycles
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Number analyzed (Participants) | 1317 | 222 | 207
Number analyzed (Cycles) | 5575 | 1021 | 2082
Days | 70.9 (41.3) | 67.6 (39.1) | 28.8 (10.8)

ADVERSE EVENTS:
Arm/Group | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300)
Serious Adverse Events (participants affected / at risk) | 12/1406 | 6/232 | 2/226
Other Adverse Events (participants affected / at risk) | 330/1406 | 68/232 | 65/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) (N=1406) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) (N=232) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300) (N=226)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flexible (Extended) Regimen no. 1 of EE20/DRSP (BAY86-5300) (N=1406) | Flexible (Extended) Regimen no. 2 of EE20/DRSP (BAY86-5300) (N=232) | Conventional Regimen of EE20/DRSP (YAZ, BAY86-5300) (N=226)
Nasopharyngitis (Infections and infestations) | 83 (95) | 15 (17) | 13 (18)
Sinusitis (Infections and infestations) | 88 (103) | 16 (17) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 93 (102) | 23 (25) | 27 (31)
Cervical dysplasia (Reproductive system and breast disorders) | 105 (112) | 21 (22) | 23 (28)

LIMITATIONS AND CAVEATS:
The Flexible (extended) Regimen no. 1 Group was enrolled under slightly different eligibility criteria for age, BMI, and fertility status than the other two treatment groups. This did not affect the results or interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of subgroup data and single center data shall not be performed until the complete study has been published. All relevant aspects regarding publication will be part of the contract between the sponsor and the investigator/institution.